CLINICAL TRIAL: NCT06163287
Title: The Effects of Drinking Hydrogen-rich Water for 6 Weeks on Exercise-related Biomarkers in Men and Women Over 50 Years Following Resistance Training Program: a Randomized Controlled Pilot Trial
Brief Title: Hydrogen-Rich Water and Exercise-Related Biomarkers in Men and Women Over 50 Years
Acronym: HYDRORES
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Novi Sad, Faculty of Sport and Physical Education (Other)
Responsible Party: Principal Investigator, Sergej Ostojic, Professor, University of Novi Sad, Faculty of Sport and Physical Education
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: HRW-1-23-AL
Record Dates: First submitted 2023-11-30; First posted 2023-12-08 (Actual); Last update posted 2024-12-04 (Actual); Status verified 2024-12

CONDITIONS: Aging
MeSH Terms: interventions — Dietary Supplements

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Supplement (Experimental): One tablet of hydrogen-rich supplement before breakfast and dinner
  Interventions: Dietary Supplement: Supplement
- Placebo (Placebo Comparator): One tablet of hydrogen-free supplement before breakfast and dinner
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Supplement — Dietary supplement containing molecular hydrogen
  Arms: Supplement
Dietary Supplement: Placebo — Inert substance
  Arms: Placebo

SUMMARY:
The study investigates the impact of consuming hydrogen-rich water over a six-week period on exercise-related biomarkers among individuals aged over 50, both men and women, who undergo a resistance training program. This research aims to discern the potential benefits of hydrogen-infused water consumption concerning exercise-related markers in an aging demographic post-resistance training.

ELIGIBILITY:
Inclusion Criteria:

* Age 50 - 65 years (at least 50% would be over 60 years)
* Body mass index 18.5 - 29.9 kg/m2
* Free of major chronic diseases or acute disorders
* Resistance exercise naïve (no resistance traiing during 6 months before study commences)

Exclusion Criteria:

* History of dietary supplement use during the 4 weeks before study commences
* Unwillingness to return for follow-up analysis

Ages: 50 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2023-10-01 (Actual); Primary Completion 2024-03-31 (Actual); Study Completion 2024-03-31 (Actual)

PRIMARY OUTCOMES:
36-Item Short Form Health Survey | Change from baseline 36-Item Short Form Health Survey total score at 6 weeks
  Short Form Health Survey total score, minimum and maximum possible score of between 0 and 100, with higher scores mean better outcome

SECONDARY OUTCOMES:
Grip strength | Change from baseline grip strength at 6 weeks
  Muscular strength generated by one's forearm muscles
Myoglobin | Change from baseline serum myoglobine at 6 weeks
  Level of myoglobin in serum
Pittsburgh Sleep Quality Index | Change from baseline Pittsburgh Sleep Quality Index score at 6 weeks
  Pittsburgh Sleep Quality Index score, a score ranging from 0 to 3, with 3 indicating the greatest dysfunction
Dehydroepiandrosterone | Change from baseline serum dehydroepiandrosterone at 6 weeks
  Level of dehydroepiandrosterone in serum

CONTACTS AND LOCATIONS:
Overall Officials: Sergej Ostojic, MD, PhD, Principal Investigator — University of Novi Sad
Locations (1):
- FSPE Applied Bioenergetics Lab, Novi Sad, Vojvodina, Serbia

IPD SHARING:
Plan to Share IPD: Yes
Data obtained through this study may be provided to qualified researchers with academic interest in hydrogen research in biomedicine. Data will be coded, with no PHI included. Approval of the request and execution of all applicable agreements are prerequisites to the sharing of data with the requesting party.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code

REFERENCES:
- [Background] Zanini D, Todorovic N, Korovljev D, Stajer V, Ostojic J, Purac J, Kojic D, Vukasinovic E, Djordjievski S, Sopic M, Guzonjic A, Ninic A, Erceg S, Ostojic SM. The effects of 6-month hydrogen-rich water intake on molecular and phenotypic biomarkers of aging in older adults aged 70 years and over: A randomized controlled pilot trial. Exp Gerontol. 2021 Nov;155:111574. doi: 10.1016/j.exger.2021.111574. Epub 2021 Oct 1. PMID 34601077
- [Background] Korovljev D, Trivic T, Drid P, Ostojic SM. Molecular hydrogen affects body composition, metabolic profiles, and mitochondrial function in middle-aged overweight women. Ir J Med Sci. 2018 Feb;187(1):85-89. doi: 10.1007/s11845-017-1638-4. Epub 2017 May 30. PMID 28560519
- [Background] Korovljev D, Stajer V, Javorac D, Ostojic SM. Hydrogen inhalation positively affects cardiometabolic risk factors in men and women aged 65 years or older: a preliminary report. Eur Geriatr Med. 2018 Oct;9(5):729-730. doi: 10.1007/s41999-018-0087-6. Epub 2018 Jul 31. No abstract available. PMID 34654221